CLINICAL TRIAL: NCT07076602
Title: Relation Between Kinematic Gait Parameters and Energy Expenditure in Children With Unilateral Lower Limb Amputation
Brief Title: Gait and Energy Expenditure in Children With Lower Limb Amputation (MAPEDE)
Acronym: MAPEDE
Status: Not yet recruiting | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC23_9872_MAPEDE; 2024-A01990-47 (Registry Identifier: ID-RCB_ANSM)
Record Dates: First submitted 2025-06-30; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Amputation of Lower Extremity, All Causes
Keywords: Children; gait analysis; energy expenditure; oxygen consumption; lower extremity amputation; kinematic; psychometry
MeSH Terms: interventions — Gait; Energy Metabolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gait and energy expenditure: Inclusion of a single day comprising two sessions of 2.5 hours each (both sessions can be interchanged) SESSION 1 : Physiotherapy assessment + Measurement of energy expenditure SESSION 2 : Measurement of kinematic parameters by gait analysis + Measurement of energy expenditure
  Interventions: Other: Gait and energy expenditure

INTERVENTIONS:
Other: Gait and energy expenditure — SESSION 1:
  Physiotherapy assessment: clinical parameters, length of limb segments, range of motion of the lower limbs, muscle strength of each lower limb joint and trunk.
  Measurement of energy expenditure:
  6-minute walking test with prosthesis, at a constant submaximal speed, with portable gas exchange analyzer to measure oxygen consumption and a connected device to calculate the Physiological Cost Index.
  * During test: recording of heart rate at the start, each minute, at the end then 5 minutes after the end, recording of the effort perceived by the child each minute (Borg scale)
  * At the end : questionnaire to assess child level of acceptability regarding the measurement of the O2 (Oxygen) consumption
  SESSION 2:
  Measurement of kinematic parameters by gait analysis: the child will be requested to walk with their prosthesis and shoes at spontaneous speed and at maximal gait speed.
  The second measurement of energy expenditure will be conducted using the same procedure as the first.

SUMMARY:
In lower limb amputation, prosthetic gait has been shown to be particularly energy-intensive. While energy expenditure has been the focus of many studies in adult amputees, this area of research is less developed for paediatric amputees. However, the increase in energy expenditure has implications for the physical, gait, and balance abilities of amputees of all ages. Combined with physical deconditioning, it exposes the patient to a greater risk of a sedentary lifestyle and weight gain, which is detrimental to their prosthetic training, autonomy, and length of hospital stay. However, this increased expenditure and deconditioning is not currently the subject of systematic evaluation in routine clinical practice for this population. In contrast to adults, the gait pattern of children amputees is poorly described, and the relation between energy expenditure and gait is rarely discussed. Oxygen consumption is the most widely used outcome to assess energy expenditure in studies. The main aim of this study was to identify the kinematic gait parameters obtained by quantified gait analysis associated with oxygen consumption during a 6-minute test in children with lower-limb amputations aged 7 years or older. This study also makes it possible to evaluate with the child's physician and rehabilitators the usefulness of measuring energy expenditure to guide medical decisions and rehabilitative care. Finally, it will allow the validation of a tool for this population for measuring energy expenditure that has been presented as more easily applicable in clinical routine than the measurement of oxygen consumption, the Physiological Cost Index (PCI). The validity and reliability of the PCI will therefore be evaluated. This study will therefore facilitate the assessment and monitoring of child amputees and provide guidance for the provision of an evidence-based rehabilitation program.

DETAILED DESCRIPTION:
The selection of subjects is carried out by the doctor of the center to which the child is attached. After obtaining consent, the study will be conducted in the movement analysis laboratory of the recruiting center, over the course of one day, comprising two sessions of 2.5 hours each. This study visit is separate from routine follow-up care.

One session will include a physiotherapy assessment and the evaluation of energy expenditure (oxygen consumption and Physiological Cost Index PCI) during a of 6-minute walking test.

The other session will include the assessment of kinematic parameters during a gait analysis and again the assessment of energy expenditure during a of 6-minute walking test.

FOLLOW-UP VISIT The report of all tests carried out will be made available to the child's physician and physiotherapists. An electronic questionnaire will be sent to them three to six months following the child' inclusion, to assess the usefulness of the information provided by the energy expenditure measurement and gait analysis in their practice.

ELIGIBILITY:
Inclusion Criteria:

* Minor aged 7 and over
* Congenital (transverse agenesis with break in limb continuity) or acquired (any etiology) transfemoral or transtibial amputation. [In the case of femoral agenesis, the flexion axis of the prosthetic knee must coincide with the contralateral one to optimize the analysis of the kinematic parameters of gait].
* Definitive prosthesis in place (no restriction on choice of prosthetic components)
* Legal representatives not opposing participation in the study for the child

Exclusion Criteria:

* Revision surgery on the residual limb within the last 3 months
* Progressive pathology associated with amputation (unstabilized sarcoma for example) which can strongly influence walking and/or energy expenditure
* Patient already included in an interventional research protocol that could lead to bias in the present study

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be drawn from the active caseload of pediatric patients with limb amputation who are currently under regular follow-up at the participating centers. These patients are monitored as part of routine clinical care. Only those meeting the predefined eligibility criteria (outlined elsewhere in the record) will be considered for inclusion. As such, the study population will reflect children and adolescents with limb amputation managed in specialized healthcare settings.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Identification of oxygen cost of walking in children with lower limb amputation | Day 1
  Oxygen cost of walking (mL.kg-1.m-1): ratio of oxygen flow rate (mL.kg-1.s-1) and walking speed (m.s-1) during 6-minute walking test. Oxygen flow rate is computed as the difference in oxygen concentration between inhaled and exhaled air during a breath. It is measured per breath and averaged over a 6-minute walking test.
Identification of gait parameters in children with lower limb amputation | Day 1
  Gait parameters are defined by :
  * deviation from a healthy pediatric norm available in the gait analysis software averaged over the entire gait cycle, calculated for the trunk, pelvis, hips, knees and ankles in each plane of space
  * deviation of center of gravity position relative to theorical position at constant speed. Spatiotemporal parameters include : speed, cadence, step length (on both sides) and stride width.

SECONDARY OUTCOMES:
Identification of the determinants of oxygen cost of walking among clinical parameters of the children with lower limb amputation | Day 1
  Oxygen cost of walking (mL.kg-1.m-1) : ratio of oxygen flow rate (mL.kg-1.s-1) and walking speed (m.s-1) during 6-minute walking test. Oxygen flow rate is computed as the difference in oxygen concentration between inhaled and exhaled air during a breath. It is measured per breath and averaged over a 6-minute walking test.
  Clinical parameters : age, sex, height, weight, level and age of amputation.
Perceived effort of the procedure for measuring oxygen consumption during the walking test assessed by the modified Borg scale | Day 1
  Modified Borg Rating of perceived exertion scales: the minimum score is 6 meaning very, very light effort, the maximum score is 10 indicating the maximum exertion.
Acceptability of the procedure for measuring the children's oxygen consumption when walking assessed by a self-questionnaire | Day 1
  This self-questionnaire designed for the study consists of 4 questions with 5 answers to assess the degree of acceptability.
  The questions are :
  * During the test, did you find the sensations associated with the MASK unpleasant?
  * Did you find the sensations associated with the DEVICE (COSMED) unpleasant?
  * Did you feel comfortable and well supported by the examiner during the test?
  * Would you be willing to take this test again if we offered it to you?
Usefulness of informations provided by the energy expenditure measurement and gait analysis assessed by a self-questionnaire | from 3 to 6 months post-inclusion
  This self-questionnaire named "Assessment of the study's clinical impact" and specially designed for the study will be addressed to the child's physician, physiotherapist or/and orthoprosthetist of the children amputees to assess the impact of energy expenditure measurement and gait analysis in guiding medical decisions and rehabilitative care at three to six months post enrolment. This self-questionnaire does not have an associated score.
Validation of the Physiological Cost Index (PCI) for the energy expenditure analysis in clinical routine | Day 1 / Session 1 and Session 2
  PCI formula : "PCI (beat/m) = [end Hearth Rate (HR) - Rest HR (beat/min)] / walking speed at the last minute of the 6 minutes walking test (m/min)"

CONTACTS AND LOCATIONS:
Overall Officials: LAURANE MAIGNAN-GOTER, Principal Investigator — Centre 01 - CHU de RENNES, Hôpital Pontchaillou
Locations (5):
- France (5):
  - Centre 02 - CHU Brest, Hôpital Morvan, Brest
  - Centre 04 - Hospices Civils de Lyon, Hôpital Mère Enfant Groupement Hospitalier Est, Bron
  - Centre 03 - CHU Dijon, Hôpital Le Bocage, Dijon
  - Centre 01 - CHU de RENNES, Hôpital Pontchaillou, Rennes
  - Hôpitaux Paris Est Val-de-Marne, Hôpital Saint-Maurice, Saint-Maurice

IPD SHARING:
Plan to Share IPD: No